CLINICAL TRIAL: NCT06958562
Title: Relation Between Lymphocyte-to-C-Reactive Protein Ratio and Coronary Artery Disease Complexity
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alsayed Ali Mahmoud Ahmed, Principal investigator, Department of cardiology, Assiut University, Assiut University
Other Study IDs: LCR ratio and CAD complexity
Record Dates: First submitted 2025-04-12; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Lymphocyte Count

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- STEMI patients undergoing primary PCI: Description: Patients diagnosed with ST-segment elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PCI) within 12 hours of symptom onset.
  Interventions: Diagnostic Test: No intervention administered. Standard care will be provided. Blood samples for lymphocyte count and CRP will be collected, and Syntax score will be calculated from angiography.
- Elective PCI Patients: Description: Patients undergoing elective coronary angiography and PCI for stable coronary artery disease.
  Interventions: Diagnostic Test: No intervention administered. Standard care will be provided. Blood samples for lymphocyte count and CRP will be collected, and Syntax score will be calculated from angiography.

INTERVENTIONS:
Diagnostic Test: No intervention administered. Standard care will be provided. Blood samples for lymphocyte count and CRP will be collected, and Syntax score will be calculated from angiography. — No intervention administered. Standard care will be provided. Blood samples for lymphocyte count and CRP will be collected, and Syntax score will be calculated from angiography.

SUMMARY:
Aim(s) of the Research :

1. To assess the relationship between the lymphocyte-to-CRP ratio and CAD complexity as assessed by Syntax score in both emergency (STEMI patients undergoing PPCI) and elective settings (patients undergoing scheduled CA plus PCI).
2. To test the relation between the LCR ratio and short-term major adverse cardiac events (MACE) within 6 months duration in patient undergoing primary PCI.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) remain the leading cause of mortality globally, responsible for approximately 17.9 million deaths annually, with over 75% occurring in low- and middle-income countries . Coronary artery disease (CAD is the leading contributor to cardiovascular-related deaths. It accounts for 45% of total fatalities linked to cardiovascular conditions .

ST-segment elevation myocardial infarction (STEMI), a severe manifestation of coronary artery disease (CAD), is a medical emergency requiring immediate revascularization to prevent irreversible myocardial damage and reduce mortality .

Primary percutaneous coronary intervention (PCI) is the preferred reperfusion strategy for STEMI, significantly reducing mortality and major adverse cardiovascular events (MACE) compared to fibrinolysis . The complexity of coronary lesions during PCI is quantified using the Syntax score, an angiographic tool that predicts procedural success and long-term outcomes . A higher Syntax score indicates increased lesion complexity, worse prognosis, and a greater risk of complications, including arrhythmias, cardiogenic shock, and heart failure .

Vascular inflammation is a key factor in the onset, progression, plaque instability, and eventual rupture of atherosclerosis . As a result, numerous inflammatory biomarkers have gained significant interest.

The inflammatory process begins with the infiltration of inflammatory cells and plays a central role in atherosclerosis, starting from its earliest stages. As atherosclerosis progresses, inflammation has been strongly associated with strokes and acute myocardial infarctions (MI) .

Systemic inflammation plays a pivotal role in the pathophysiology of atherosclerosis and its complications . Inflammatory markers, such as elevated C-reactive protein (CRP), have been shown to predict adverse outcomes in CAD . Concurrently, lymphopenia is a marker of immune suppression and poor cardiovascular prognosis .

C-reactive protein (CRP) is a well-established marker of inflammation commonly used to monitor infections and inflammatory disorders. Lymphocytes, as key players in the immune response, tend to decrease in number during excessive immune activation . In clinical practice, markers such as leukocytes, neutrophils, lymphocytes, platelets, and CRP are routinely measured as indicators of inflammation. Combining these biomarkers may provide greater reliability and diagnostic accuracy than relying on a single marker alone.

The lymphocyte-to-CRP (LCR) ratio, which combines these two markers, has emerged as a promising biomarker for risk stratification in acute coronary syndromes .

The C-reactive protein-to-lymphocyte ratio (CLR) has emerged as a novel inflammatory biomarker, offering potential for predicting prognosis and aiding in the diagnostic evaluation of various conditions. For instance, elevated CLR levels have been associated with poor outcomes in COVID-19 patients , as well as in those with severe fever and thrombocytopenia syndrome . Additionally, high CLR levels have been linked to unfavorable prognoses in patients with malignant diseases . Despite this growing evidence, the relationship between CLR and MI remains underexplored.

Preliminary studies suggest that a lower LCR ratio is associated with increased CAD severity and poorer outcomes . However, the relationship between LCR ratio and Syntax score, particularly in STEMI patients undergoing primary PCI, remains underexplored. Similarly, its relevance in elective PCI, where lesion complexity and systemic inflammation may differ, has not been fully investigated.

While both Syntax score and LCR ratio provide valuable prognostic information, there is limited evidence on their interplay and predictive value for short-term outcomes in STEMI and elective PCI patients. By addressing this gap, this study aims to improve risk stratification and clinical decision-making .

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 to 80 years

Diagnosed with STEMI undergoing primary PCI within 12 hours of symptom onset

Patients undergoing elective PCI with documented coronary artery disease

Provided written informed consent

Exclusion Criteria:

Previous history of myocardial infarction, PCI, or coronary artery bypass grafting (CABG)

Diagnosed autoimmune or chronic inflammatory disorders

Active infection or malignancy at the time of presentation

Severe renal impairment (eGFR <30 mL/min/1.73 m²) or hepatic dysfunction

Use of immunosuppressive therapy

Diagnosis of acute or chronic leukemia within the past 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-06-03 (Estimated); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Relationship between Lymphocyte-to-CRP ratio and CAD complexity assessed by Syntax score | At baseline during coronary angiography
  To assess the correlation between the lymphocyte-to-C-reactive protein (LCR) ratio and coronary artery disease (CAD) complexity as measured by Syntax score in STEMI and elective PCI patients.

SECONDARY OUTCOMES:
Association between Lymphocyte-to-CRP ratio and short-term major adverse cardiac events (MACE) | Within 3 months after PCI
  To evaluate the association between the LCR ratio and the incidence of major adverse cardiac events (MACE) within 6 months in patients undergoing primary PCI.

IPD SHARING:
Plan to Share IPD: Undecided